CLINICAL TRIAL: NCT06214611
Title: Adaptive Radiotherapy in the Treatment of Patients With a Histologically Confirmed Malignant Tumor in the Head and Neck Region: Prospective Validation of ART in Patients With HNT (Prospektive Validierung Der ART Bei Patientinnen Und Patienen Mit Kopf-Hals Tumoren,)
Brief Title: Prospective Validation of Adaptive Radiotherapy (ART) in Patients With Head and Neck Tumors
Acronym: ART in HNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Maja Guberina, PD Dr. med. (MD) Maja Guberina, specialist in radiation oncology, senior consultant, University Hospital, Essen
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-11129-BO; DRKS00033144 (Other: DRKS, Deutsches Register Klinischer Studien)
Record Dates: First submitted 2023-12-28; First posted 2024-01-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Cancer; Adaptive Radiotherapy; Radiation; Optimized Treatment; Protection of Organs at Risk; Dysphagia Reduction
Keywords: Head and Neck Cancer; Adaptive Radiotherapy; Protection of organs at risk; Optimized treatment; Dysphagia reduction
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Adaptive Radiotherapy (Other): Adaptive Radiation Therapy
  Interventions: Radiation: Adaptive Radiotherapy
- Standard Treatment Arm, IGRT (Active Comparator): Standard Treatment Arm, IGRT
  Interventions: Radiation: Adaptive Radiotherapy

INTERVENTIONS:
Radiation: Adaptive Radiotherapy — Adaptive Radiotherapy in the head and neck region
  Other Names: Dysphagia optimized Adaptive Radiotherapy (ART)

SUMMARY:
Adaptive radiotherapy (ART) includes image-guided radiotherapy (IGRT) and also offers further possibilities for plan adaptation. A particularly high benefit can be expected for patients in whom the clinical target volume (CTV) can show a significant change in shape from fraction to fraction due to anatomical deviations. The shape and position constancy of the CTV during the course of the series is examined in this trial. Dosimetric disadvantages of this type have not been reported so far. The aim of this study is to identify patients who benefit from ART at an early stage and to select them for this method, and then to continue to offer ART to this patient group. If a relevant reduction in the minimum planning target volume (PTV) margins with ART compared to IGRT is demonstrated in this study, patients could be treated with ART.

DETAILED DESCRIPTION:
The aim here is to prospectively evaluate modern technical standards. In the last 25 years, radiotherapy has developed rapidly away from two-dimensional procedures towards volume-modulated, three-dimensional techniques. But here, too, there is a broad radiotherapeutic spectrum due to the high technical diversity in radiotherapy and ever newer technical innovations. (1) Definitive radiochemotherapy is standard of care for locally advanced head and neck tumors. The aim of this study is to monitor the influence of the new technical therapy standards (therapy options in application: volume-modulated rapid-arc technique (VMAT) / online onboard image-guidance (IGRT) and adaptive re-planning, using the linear accelerator ETHOS currently established and installed at the Department of Radiotherapy in December 2021) as a function of dose parameters for quality assurance of feasibility.

Therapy with ETHOS represents a comprehensive new treatment option that is tailored and individualized from the initial planning and adjustment on the treatment table to radiation monitoring of the whole therapy.

Online-adaptive radiotherapy (ART) allows the dose distribution to be adapted to the anatomical changes online and immediately before each radiation fraction. Adaptive radiotherapy is a further development of image-guided radiotherapy (IGRT), which is now standard of care in radiotherapy. In contrast to ART, with IGRT the radiation plan cannot be adapted to deformations of the body from radiation fraction to radiation fraction, e.g. through different positioning of the tongue or jaw.

This trial creates the basis for standardizing treatment parameters as far as possible, but also for introducing improvements in the treatment of future patients in a personalized and individualized form.

Standard therapy can be further optimized using modern equipment and high-precision linear accelerators.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG 0-1
2. Histopathology confirmation
3. Compliance
4. Tumor in the head and neck region
5. Indication for radiotherapy

Exclusion Criteria:

1. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Accumulated dose distribution in CTV | 2 weeks
  accumulated dose distribution in the clinical target volume, EUD [Gy]

SECONDARY OUTCOMES:
dysphagia assessment scores | 2 weeks to 5 years
  dysphagia assessment scores
Minimally isotropic PTV margin | 2 months
  Minimally isotropic PTV margin [mm]
Progression free survival (PFS) | 2 months to 5 years
  Progression free survival (PFS)
overall survival (OS) | 2 months to 5 years
  overall survival (OS)
dose organs at risk (OAR) | 2 weeks
  dose organs at risk (OAR)
Side effects, LENT-SOMA | 2 months to 5 years
  LENT-SOMA criteria and score for Adverse Events (CTCAE)
quality of life (EORTC) | 2 months to 5 years
  quality of life (EORTC)
Side effects (CTC AE) | 2 months to 5 years
  Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Radiotherapy, University Hospital Essen, National Center for Tumor Diseases (NCT) West, Essen, Germany / NRW, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chetty IJ, Martel MK, Jaffray DA, Benedict SH, Hahn SM, Berbeco R, Deye J, Jeraj R, Kavanagh B, Krishnan S, Lee N, Low DA, Mankoff D, Marks LB, Ollendorf D, Paganetti H, Ross B, Siochi RA, Timmerman RD, Wong JW. Technology for Innovation in Radiation Oncology. Int J Radiat Oncol Biol Phys. 2015 Nov 1;93(3):485-92. doi: 10.1016/j.ijrobp.2015.07.007. Epub 2015 Jul 11. PMID 26460989